CLINICAL TRIAL: NCT06208644
Title: Identification of Obstacles and Levers to Interdisciplinary Work in Palliative Care Units
Acronym: Work-in-PCU
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9027
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-01

CONDITIONS: Palliative Care
Keywords: Palliative Care; Palliative Care Units

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Palliative care is active care delivered by a multidisciplinary team, in a global approach to the person suffering from a serious, progressive illness, in an advanced phase, with a fatal outcome. Their goal is to relieve physical pain and other symptoms, but also to take into account psychological, social and spiritual suffering.

Palliative care and support are interdisciplinary. They are aimed at the patient as an individual, their family and loved ones, at home or in an institution. Training and support for caregivers and volunteers are part of this approach.

Recent years have seen the development of teaching in the discipline both during the initial course and through continuing training actions, the latter based on the very notion of multi-professionality. But it is clear that during the initial course of health professionals, learning remains confined to professions, in silos.

It is in view of this observation that the 2015-2018 palliative care development plan in France proposed the establishment of transversal teaching, for health students, through its measures 4.1 and 4.2, lessons put in place at through local initiatives which are still underdeveloped.

It is therefore appropriate to question the methods of learning "know how to work together". This work therefore aims to reflect, through what can promote but also hinder interdisciplinary work, on the way in which health students can be taught to work in interdisciplinarity and in particular during their internships in palliative care structures

ELIGIBILITY:
Inclusion Criteria:

* Health professionals, all professions combined, working in palliative care units agreeing to participate in research
* Health students (hospital students, nurses, etc.) doing an internship in a palliative care unit agreeing to participate in research
* Agreeing to participate in the study

Exclusion Criteria:

* Refusal to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health professionals working in palliative care unit and Health students (hospital students, nurses, etc.) doing an internship in this unit.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Review of the perception of interdisciplinarity and interdisciplinary work among staff working or doing an internship in a palliative care unit | Study covers the period from August 25, 2023 to October 25, 2023
  The study consisted of an inventory of the perception of interdisciplinarity and interdisciplinary work among staff working or doing an internship in a palliative care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Service de soins Palliatifs - CHU de Strasbourg - France, Strasbourg, France